CLINICAL TRIAL: NCT05065684
Title: Effect of rhBMP-2 or rhBMP-7 on Long Bone Fractures and Non-unions.
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: Effect of rhBMP-2 or rhBMP-7
Record Dates: First submitted 2021-09-13; First posted 2021-10-04 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2021-08

CONDITIONS: Long Bone Non-union
Keywords: Long bone non-union

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rhBMP-2 and rhBMP-7: patients who have been treated with rhBMP-2 or rhBMP-7 for long bone non-union or acute fractures
- No-BMP: patients who have been treated with standart care, i.e. non-union resection and autologous bone graft

SUMMARY:
Delayed fracture healing continues to cause significant patient morbidity and economic burden to society. Biological stimulation of acute fractures and non-unions includes application of rhBMP-2 and rhBMP-7. However, BMP use continues to be a matter of controversy as literature shows scarce evidence for treatment effectiveness. The aim of this study is to compare acute fractures and non-unions in the long bones humerus, femur and tibia with and without BMP treatment of acute fractures. Furthermore, the investigators want to identify complications and risk factors on union-rate and time to union.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective is to assess time to union and union rate after rhBMP-2 and rhBMP-7 application at long bone fractures and non-unions.

Secondary Objective(s):

* Analysis of secondary complications
* Analysis of risk factors

Hypothesis and Statistical considerations and estimated enrollment:

The investigators hypothesize that with the use of rhBMP-2 and rhBMP-7 there will be a faster timer to union and higher union rate compared to no-BMP. Outcomes will be assessed prospectively.

This study is exploratory in nature. Therefore, there is no formal statistical hypothesis and no formal sample size calculation. Approximately 150 long-bone fractures and non-unions are expected.

Data will be analyzed with the use of simple summary statistics. Depending on the volume and quality of the collected data, different statistical analyses will be applied. Exploratory analyses will be conducted to investigate relationships between the different treatment options and the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Long bone fracture or long bone non-union.
* Signed informed consent, if required by IRB/EC

Exclusion Criteria:

Prisoner at date of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute fracture or non-union of a long-bone
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time to Union | 24 months
  Time to Union in months
Union-rate | 24 months
  Union-rate in percentage

SECONDARY OUTCOMES:
Risk factor analysis | 24 months
  Clinically relevant retrospective data regarding medical history, co-morbidity, the localization and the outcome will be collected. Comorbidities are listed and categorized as follows: Cardiovascular (peripheral arterial disease, hyperuricemia, coronary artery disease, bleeding disorders, hemophilia A, thrombocytopenia, blood loss anemia), metabolic (diabetes, adiposities, hypertonia, metabolic syndrome, liver disorders, alcoholic liver cirrhosis, alcohol abuse, hypothyroidism, hyperkalemia), neurologic (Parkinson, borderline personality, suicidality, epilepsy, drug abuse, sleep apnea syndrome, status post apoplexy), rheumatologic and allergic (atopic eczema, rheumatoid arthritis, bronchial asthma, chronic bronchitis) and infectious (MRSA, hepatitis A, B and C).
complications/Adverse Events related to implant or surgery | 24 months
  complications/Adverse Events related to implant or surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Raschke, Prof. Dr., Principal Investigator — University Hospital Muenster

IPD SHARING:
Plan to Share IPD: No